CLINICAL TRIAL: NCT06857136
Title: The Role of the Glymphatic System Avaluated Thourgh mr Imaging in the Diagnosis and Management of NPH
Acronym: GLINFANPH_2021
Status: Completed | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: GLINFANPH_2021
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-02

CONDITIONS: Hydrocephalus; Normal Pressure Hydrocephalus
Keywords: hydrocephalus; Normal pressure hydrocephalus; NPH; Glymphatic System; DTI-ALPS; Diffusion Tensor Imaging; ALPS-index
MeSH Terms: conditions — Hydrocephalus; Hydrocephalus, Normal Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients attending the NPH outpatient clinic were prospectively enrolled in the study. The inclusion criteria were: (i) clinical and radiological diagnosis of probable NPH according to existing guidelines and (ii) age of over 50 years. Exclusion criteria were: (i) inability to undergo MR; (ii) a diagnosis of any other neurological pathology, particularly neurodegenerative or neuroinflammatory; (iii) previous neurosurgical interventions on the brain of any type; (iv) inability to undergo general anaesthesia.
- Control group: A healthy control group of patients (HC group) matched for age with the IR group, underwent MR with DTI-ALPS study. Exclusion criteria for this group were: (i) a previous diagnosis of any neurological disorder of any type. (ii) a history of neurosurgical intervention of any kind; and (iii) a prior diagnosis of malignancy of any type.

SUMMARY:
The goal of this observational study is to evaluate the role of DTI-ALPS in the diagnostic and therapeutic management of NPH

The main questions it aims to answer are:

* Whether the glymphatic system (GS) is actually impaired in NPH
* Whether DTI-ALPS index can predict the positive response to tap test (TT) and to ventriculo-peritoneal shunt (VPS) surgery.

A healthy control group of patients (HC group) matched for age with the study group, will undergo MR with DTI-ALPS study

DETAILED DESCRIPTION:
Enrolled patients followed a diagnostic-therapeutic pathway, consisting of the following steps:

* t0: MR with DTI-ALPS study;
* t1 (within 7 days from T0): clinical and neurosurgical assessment with NPH-specific rating scales (detailed below) before and after a lumbar TT, including measurements of opening pressure, drainage of 40-50 mL of CSF and collection of samples for neurodegenerative biomarkers (β-Amyloid 40, 42 total and P-Tau) quantification. An MR with DTI-ALPS study within 6 hours from TT;
* t2 (within 3 months from T1): patients with a positive TT response (included responders, IR group) underwent VPS surgery, with CSF samples collected for the same neurodegenerative biomarkers (β-Amyloid 40, 42 total and P-Tau);
* t3 (three months after surgery, IR group only): clinical and neurosurgical evaluation using NPH-specific rating scales to classify patients as improved, unchanged, or worsened compared to their preoperative condition; MR with DTI-ALPS study.

ELIGIBILITY:
Suspected NPH patients according to the following:

Inclusion Criteria:

* clinical and radiological diagnosis of probable NPH according to existing guidelines
* age of over 50 years

Exclusion Criteria:

* inability to undergo MR
* diagnosis of any other neurological pathology, particularly neurodegenerative or neuroinflammatory
* previous neurosurgical interventions on the brain of any type.
* inability to undergo general anaesthesia

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients affected by normal pressure hydrocephalus
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison between study and control group | 4 years
  Difference in DTI ALPS index between NPH patients and healthy controls

SECONDARY OUTCOMES:
Difference in response to tap test between NPH patients who responded and those who did not | 4 years
  Difference in DTI ALPS index between NPH who responded to tap test (and underwent to ventircolopetoneal shunt) and those who did not
Change in DTI ALPS index across treatment in NPH patients | 4 years
  Difference in DTI ALPS index in NPH patients between T0 (before TT), T1 (after TT) and T3 (after VP shunt)
Change in CSF degenerative biomarker concentrations | 4 years
  CSF degenerative biomarkers (total tau protein, p-181 tau protein, Aβ42 e Aβ40 protein) variation between T1, T2 and T3

CONTACTS AND LOCATIONS:
Overall Officials: Morgan A Broggi, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abu-Rumeileh S, Giannini G, Polischi B, Albini-Riccioli L, Milletti D, Oppi F, Stanzani-Maserati M, Capellari S, Mantovani P, Palandri G, Cortelli P, Cevoli S, Parchi P. Revisiting the Cerebrospinal Fluid Biomarker Profile in Idiopathic Normal Pressure Hydrocephalus: The Bologna Pro-Hydro Study. J Alzheimers Dis. 2019;68(2):723-733. doi: 10.3233/JAD-181012. PMID 30883350
- [Background] Graff-Radford NR. Alzheimer CSF biomarkers may be misleading in normal-pressure hydrocephalus. Neurology. 2014 Oct 21;83(17):1573-5. doi: 10.1212/WNL.0000000000000916. PMID 25332445
- [Background] Appollonio I, Leone M, Isella V, Piamarta F, Consoli T, Villa ML, Forapani E, Russo A, Nichelli P. The Frontal Assessment Battery (FAB): normative values in an Italian population sample. Neurol Sci. 2005 Jun;26(2):108-16. doi: 10.1007/s10072-005-0443-4. PMID 15995827
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Tinetti ME, Williams TF, Mayewski R. Fall risk index for elderly patients based on number of chronic disabilities. Am J Med. 1986 Mar;80(3):429-34. doi: 10.1016/0002-9343(86)90717-5. PMID 3953620
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Tian Y, Cai X, Zhou Y, Jin A, Wang S, Yang Y, Mei L, Jing J, Li S, Meng X, Wei T, Liu T, Wang Y, Pan Y, Wang Y. Impaired glymphatic system as evidenced by low diffusivity along perivascular spaces is associated with cerebral small vessel disease: a population-based study. Stroke Vasc Neurol. 2023 Oct;8(5):413-423. doi: 10.1136/svn-2022-002191. Epub 2023 Apr 12. PMID 37045543
- [Background] Shanks J, Markenroth Bloch K, Laurell K, Cesarini KG, Fahlstrom M, Larsson EM, Virhammar J. Aqueductal CSF Stroke Volume Is Increased in Patients with Idiopathic Normal Pressure Hydrocephalus and Decreases after Shunt Surgery. AJNR Am J Neuroradiol. 2019 Mar;40(3):453-459. doi: 10.3174/ajnr.A5972. Epub 2019 Feb 21. PMID 30792248
- [Background] Morone PJ, Dewan MC, Zuckerman SL, Tubbs RS, Singer RJ. Craniometrics and Ventricular Access: A Review of Kocher's, Kaufman's, Paine's, Menovksy's, Tubbs', Keen's, Frazier's, Dandy's, and Sanchez's Points. Oper Neurosurg. 2020 May 1;18(5):461-469. doi: 10.1093/ons/opz194. PMID 31420653
- [Background] Walchenbach R, Geiger E, Thomeer RT, Vanneste JA. The value of temporary external lumbar CSF drainage in predicting the outcome of shunting on normal pressure hydrocephalus. J Neurol Neurosurg Psychiatry. 2002 Apr;72(4):503-6. doi: 10.1136/jnnp.72.4.503. PMID 11909911
- [Background] Razay G, Vreugdenhil A, Liddell J. A prospective study of ventriculo-peritoneal shunting for idiopathic normal pressure hydrocephalus. J Clin Neurosci. 2009 Sep;16(9):1180-3. doi: 10.1016/j.jocn.2008.12.007. Epub 2009 Jun 3. PMID 19497748
- [Background] Toma AK, Stapleton S, Papadopoulos MC, Kitchen ND, Watkins LD. Natural history of idiopathic normal-pressure hydrocephalus. Neurosurg Rev. 2011 Oct;34(4):433-9. doi: 10.1007/s10143-011-0316-7. Epub 2011 May 19. PMID 21594683
- [Background] Andren K, Wikkelso C, Tisell M, Hellstrom P. Natural course of idiopathic normal pressure hydrocephalus. J Neurol Neurosurg Psychiatry. 2014 Jul;85(7):806-10. doi: 10.1136/jnnp-2013-306117. Epub 2013 Nov 29. PMID 24292998
- [Background] Iseki C, Kawanami T, Nagasawa H, Wada M, Koyama S, Kikuchi K, Arawaka S, Kurita K, Daimon M, Mori E, Kato T. Asymptomatic ventriculomegaly with features of idiopathic normal pressure hydrocephalus on MRI (AVIM) in the elderly: a prospective study in a Japanese population. J Neurol Sci. 2009 Feb 15;277(1-2):54-7. doi: 10.1016/j.jns.2008.10.004. Epub 2008 Nov 5. PMID 18990411
- [Background] Iseki C, Takahashi Y, Wada M, Kawanami T, Adachi M, Kato T. Incidence of idiopathic normal pressure hydrocephalus (iNPH): a 10-year follow-up study of a rural community in Japan. J Neurol Sci. 2014 Apr 15;339(1-2):108-12. doi: 10.1016/j.jns.2014.01.033. Epub 2014 Feb 3. PMID 24656600
- [Background] Fukuhara T, Luciano MG. Clinical features of late-onset idiopathic aqueductal stenosis. Surg Neurol. 2001 Mar;55(3):132-6; discussion 136-7. doi: 10.1016/s0090-3019(01)00359-7. PMID 11311904
- [Background] Ved R, Leach P, Patel C. Surgical treatment of long-standing overt ventriculomegaly in adults (LOVA). Acta Neurochir (Wien). 2017 Jan;159(1):71-79. doi: 10.1007/s00701-016-2998-7. Epub 2016 Nov 2. PMID 27807671
- [Background] Palandri G, Carretta A, La Corte E, Giannini G, Martinoni M, Mantovani P, Albini-Riccioli L, Tonon C, Mazzatenta D, Elder BD, Conti A. Open-aqueduct LOVA, LIAS, iNPH: a comparative clinical-radiological study exploring the "grey zone" between different forms of chronic adulthood hydrocephalus. Acta Neurochir (Wien). 2022 Jul;164(7):1777-1788. doi: 10.1007/s00701-022-05215-9. Epub 2022 Apr 27. PMID 35477816
- [Background] Miyamoto J, Tatsuzawa K, Inoue Y, Imahori Y, Mineura K. Oxygen metabolism changes in patients with idiopathic normal pressure hydrocephalus before and after shunting operation. Acta Neurol Scand. 2007 Sep;116(3):137-43. doi: 10.1111/j.1600-0404.2007.00798.x. PMID 17714325
- [Background] Ishii K, Hashimoto M, Hayashida K, Hashikawa K, Chang CC, Nakagawara J, Nakayama T, Mori S, Sakakibara R. A multicenter brain perfusion SPECT study evaluating idiopathic normal-pressure hydrocephalus on neurological improvement. Dement Geriatr Cogn Disord. 2011;32(1):1-10. doi: 10.1159/000328972. Epub 2011 Jul 29. PMID 21811073
- [Background] Mataro M, Matarin M, Poca MA, Pueyo R, Sahuquillo J, Barrios M, Junque C. Functional and magnetic resonance imaging correlates of corpus callosum in normal pressure hydrocephalus before and after shunting. J Neurol Neurosurg Psychiatry. 2007 Apr;78(4):395-8. doi: 10.1136/jnnp.2006.096164. Epub 2006 Oct 20. PMID 17056634
- [Background] Khoo HM, Kishima H, Tani N, Oshino S, Maruo T, Hosomi K, Yanagisawa T, Kazui H, Watanabe Y, Shimokawa T, Aso T, Kawaguchi A, Yamashita F, Saitoh Y, Yoshimine T. Default mode network connectivity in patients with idiopathic normal pressure hydrocephalus. J Neurosurg. 2016 Feb;124(2):350-8. doi: 10.3171/2015.1.JNS141633. Epub 2015 Aug 21. PMID 26295919
- [Background] Miyati T, Mase M, Kasai H, Hara M, Yamada K, Shibamoto Y, Soellinger M, Baltes C, Luechinger R. Noninvasive MRI assessment of intracranial compliance in idiopathic normal pressure hydrocephalus. J Magn Reson Imaging. 2007 Aug;26(2):274-8. doi: 10.1002/jmri.20999. PMID 17610284
- [Background] Algin O, Hakyemez B, Parlak M. The efficiency of PC-MRI in diagnosis of normal pressure hydrocephalus and prediction of shunt response. Acad Radiol. 2010 Feb;17(2):181-7. doi: 10.1016/j.acra.2009.08.011. Epub 2009 Nov 11. PMID 19910214
- [Background] Battal B, Kocaoglu M, Bulakbasi N, Husmen G, Tuba Sanal H, Tayfun C. Cerebrospinal fluid flow imaging by using phase-contrast MR technique. Br J Radiol. 2011 Aug;84(1004):758-65. doi: 10.1259/bjr/66206791. Epub 2011 May 17. PMID 21586507
- [Background] Taoka T, Ito R, Nakamichi R, Kamagata K, Sakai M, Kawai H, Nakane T, Abe T, Ichikawa K, Kikuta J, Aoki S, Naganawa S. Reproducibility of diffusion tensor image analysis along the perivascular space (DTI-ALPS) for evaluating interstitial fluid diffusivity and glymphatic function: CHanges in Alps index on Multiple conditiON acquIsition eXperiment (CHAMONIX) study. Jpn J Radiol. 2022 Feb;40(2):147-158. doi: 10.1007/s11604-021-01187-5. Epub 2021 Aug 14. PMID 34390452
- [Background] Thavarajasingam SG, El-Khatib M, Vemulapalli K, Iradukunda HAS, K SV, Borchert R, Russo S, Eide PK. Radiological predictors of shunt response in the diagnosis and treatment of idiopathic normal pressure hydrocephalus: a systematic review and meta-analysis. Acta Neurochir (Wien). 2023 Feb;165(2):369-419. doi: 10.1007/s00701-022-05402-8. Epub 2022 Nov 26. PMID 36435931
- [Background] Carlsen JF, Munch TN, Hansen AE, Hasselbalch SG, Rykkje AM. Can preoperative brain imaging features predict shunt response in idiopathic normal pressure hydrocephalus? A PRISMA review. Neuroradiology. 2022 Nov;64(11):2119-2133. doi: 10.1007/s00234-022-03021-9. Epub 2022 Jul 24. PMID 35871239
- [Background] Virhammar J, Laurell K, Cesarini KG, Larsson EM. Preoperative prognostic value of MRI findings in 108 patients with idiopathic normal pressure hydrocephalus. AJNR Am J Neuroradiol. 2014 Dec;35(12):2311-8. doi: 10.3174/ajnr.A4046. Epub 2014 Jul 10. PMID 25012669
- [Background] Virhammar J, Laurell K, Cesarini KG, Larsson EM. The callosal angle measured on MRI as a predictor of outcome in idiopathic normal-pressure hydrocephalus. J Neurosurg. 2014 Jan;120(1):178-84. doi: 10.3171/2013.8.JNS13575. Epub 2013 Sep 27. PMID 24074491
- [Background] Ishii K, Kanda T, Harada A, Miyamoto N, Kawaguchi T, Shimada K, Ohkawa S, Uemura T, Yoshikawa T, Mori E. Clinical impact of the callosal angle in the diagnosis of idiopathic normal pressure hydrocephalus. Eur Radiol. 2008 Nov;18(11):2678-83. doi: 10.1007/s00330-008-1044-4. Epub 2008 May 24. PMID 18500524
- [Background] Chen J, He W, Zhang X, Lv M, Zhou X, Yang X, Wei H, Ma H, Li H, Xia J. Value of MRI-based semi-quantitative structural neuroimaging in predicting the prognosis of patients with idiopathic normal pressure hydrocephalus after shunt surgery. Eur Radiol. 2022 Nov;32(11):7800-7810. doi: 10.1007/s00330-022-08733-3. Epub 2022 Apr 30. PMID 35501572
- [Background] Craven CL, Toma AK, Mostafa T, Patel N, Watkins LD. The predictive value of DESH for shunt responsiveness in idiopathic normal pressure hydrocephalus. J Clin Neurosci. 2016 Dec;34:294-298. doi: 10.1016/j.jocn.2016.09.004. Epub 2016 Sep 28. PMID 27692614
- [Background] Ahmed AK, Luciano M, Moghekar A, Shin J, Aygun N, Sair HI, Rigamonti D, Blitz AM. Does the Presence or Absence of DESH Predict Outcomes in Adult Hydrocephalus? AJNR Am J Neuroradiol. 2018 Nov;39(11):2022-2026. doi: 10.3174/ajnr.A5820. Epub 2018 Oct 25. PMID 30361433
- [Background] Agerskov S, Wallin M, Hellstrom P, Ziegelitz D, Wikkelso C, Tullberg M. Absence of Disproportionately Enlarged Subarachnoid Space Hydrocephalus, a Sharp Callosal Angle, or Other Morphologic MRI Markers Should Not Be Used to Exclude Patients with Idiopathic Normal Pressure Hydrocephalus from Shunt Surgery. AJNR Am J Neuroradiol. 2019 Jan;40(1):74-79. doi: 10.3174/ajnr.A5910. Epub 2018 Dec 6. PMID 30523139
- [Background] Shinoda N, Hirai O, Hori S, Mikami K, Bando T, Shimo D, Kuroyama T, Kuramoto Y, Matsumoto M, Ueno Y. Utility of MRI-based disproportionately enlarged subarachnoid space hydrocephalus scoring for predicting prognosis after surgery for idiopathic normal pressure hydrocephalus: clinical research. J Neurosurg. 2017 Dec;127(6):1436-1442. doi: 10.3171/2016.9.JNS161080. Epub 2017 Feb 3. PMID 28156249
- [Background] Halperin JJ, Kurlan R, Schwalb JM, Cusimano MD, Gronseth G, Gloss D. Practice guideline: Idiopathic normal pressure hydrocephalus: Response to shunting and predictors of response: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology. Neurology. 2015 Dec 8;85(23):2063-71. doi: 10.1212/WNL.0000000000002193. PMID 26644048
- [Background] O'Hayon BB, Drake JM, Ossip MG, Tuli S, Clarke M. Frontal and occipital horn ratio: A linear estimate of ventricular size for multiple imaging modalities in pediatric hydrocephalus. Pediatr Neurosurg. 1998 Nov;29(5):245-9. doi: 10.1159/000028730. PMID 9917541
- [Background] Eklund A, Smielewski P, Chambers I, Alperin N, Malm J, Czosnyka M, Marmarou A. Assessment of cerebrospinal fluid outflow resistance. Med Biol Eng Comput. 2007 Aug;45(8):719-35. doi: 10.1007/s11517-007-0199-5. Epub 2007 Jul 17. PMID 17634761
- [Background] Marmarou A, Bergsneider M, Klinge P, Relkin N, Black PM. The value of supplemental prognostic tests for the preoperative assessment of idiopathic normal-pressure hydrocephalus. Neurosurgery. 2005 Sep;57(3 Suppl):S17-28; discussion ii-v. doi: 10.1227/01.neu.0000168184.01002.60. PMID 16160426
- [Background] Malm J, Kristensen B, Karlsson T, Fagerlund M, Elfverson J, Ekstedt J. The predictive value of cerebrospinal fluid dynamic tests in patients with th idiopathic adult hydrocephalus syndrome. Arch Neurol. 1995 Aug;52(8):783-9. doi: 10.1001/archneur.1995.00540320059013. PMID 7639630
- [Background] Haan J, Thomeer RT. Predictive value of temporary external lumbar drainage in normal pressure hydrocephalus. Neurosurgery. 1988 Feb;22(2):388-91. doi: 10.1227/00006123-198802000-00020. PMID 3352890
- [Background] Tullberg M, Blennow K, Mansson JE, Fredman P, Tisell M, Wikkelso C. Ventricular cerebrospinal fluid neurofilament protein levels decrease in parallel with white matter pathology after shunt surgery in normal pressure hydrocephalus. Eur J Neurol. 2007 Mar;14(3):248-54. doi: 10.1111/j.1468-1331.2006.01553.x. PMID 17355543
- [Background] Blennow K, Hampel H. CSF markers for incipient Alzheimer's disease. Lancet Neurol. 2003 Oct;2(10):605-13. doi: 10.1016/s1474-4422(03)00530-1. PMID 14505582
- [Background] Tullberg M, Blennow K, Mansson JE, Fredman P, Tisell M, Wikkelso C. Cerebrospinal fluid markers before and after shunting in patients with secondary and idiopathic normal pressure hydrocephalus. Cerebrospinal Fluid Res. 2008 Apr 25;5:9. doi: 10.1186/1743-8454-5-9. PMID 18439296
- [Background] Tarnaris A, Toma AK, Kitchen ND, Watkins LD. Ongoing search for diagnostic biomarkers in idiopathic normal pressure hydrocephalus. Biomark Med. 2009 Dec;3(6):787-805. doi: 10.2217/bmm.09.37. PMID 20477715
- [Background] Patel S, Lee EB, Xie SX, Law A, Jackson EM, Arnold SE, Clark CM, Shaw LM, Grady MS, Trojanowski JQ, Hamilton RH. Phosphorylated tau/amyloid beta 1-42 ratio in ventricular cerebrospinal fluid reflects outcome in idiopathic normal pressure hydrocephalus. Fluids Barriers CNS. 2012 Mar 23;9(1):7. doi: 10.1186/2045-8118-9-7. PMID 22444461
- [Background] Li X, Miyajima M, Mineki R, Taka H, Murayama K, Arai H. Analysis of potential diagnostic biomarkers in cerebrospinal fluid of idiopathic normal pressure hydrocephalus by proteomics. Acta Neurochir (Wien). 2006 Aug;148(8):859-64; discussion 864. doi: 10.1007/s00701-006-0787-4. Epub 2006 Jun 6. PMID 16755327
- [Background] Li X, Miyajima M, Jiang C, Arai H. Expression of TGF-betas and TGF-beta type II receptor in cerebrospinal fluid of patients with idiopathic normal pressure hydrocephalus. Neurosci Lett. 2007 Feb 14;413(2):141-4. doi: 10.1016/j.neulet.2006.11.039. Epub 2006 Dec 27. PMID 17194537
- [Background] Chen Z, Liu C, Zhang J, Relkin N, Xing Y, Li Y. Cerebrospinal fluid Abeta42, t-tau, and p-tau levels in the differential diagnosis of idiopathic normal-pressure hydrocephalus: a systematic review and meta-analysis. Fluids Barriers CNS. 2017 May 10;14(1):13. doi: 10.1186/s12987-017-0062-5. PMID 28486988
- [Background] Santangelo R, Cecchetti G, Bernasconi MP, Cardamone R, Barbieri A, Pinto P, Passerini G, Scomazzoni F, Comi G, Magnani G. Cerebrospinal Fluid Amyloid-beta 42, Total Tau and Phosphorylated Tau are Low in Patients with Normal Pressure Hydrocephalus: Analogies and Differences with Alzheimer's Disease. J Alzheimers Dis. 2017;60(1):183-200. doi: 10.3233/JAD-170186. PMID 28826180
- [Background] Graff-Radford NR, Jones DT. Normal Pressure Hydrocephalus. Continuum (Minneap Minn). 2019 Feb;25(1):165-186. doi: 10.1212/CON.0000000000000689. PMID 30707192
- [Background] Bono F, Lupo MR, Serra P, Cantafio C, Lucisano A, Lavano A, Fera F, Pardatscher K, Quattrone A. Obesity does not induce abnormal CSF pressure in subjects with normal cerebral MR venography. Neurology. 2002 Nov 26;59(10):1641-3. doi: 10.1212/01.wnl.0000035628.81384.5f. PMID 12451215
- [Background] Wilson RK, Williams MA. The role of the neurologist in the longitudinal management of normal pressure hydrocephalus. Neurologist. 2010 Jul;16(4):238-48. doi: 10.1097/NRL.0b013e3181de4907. PMID 20592567
- [Background] Marmarou A, Young HF, Aygok GA, Sawauchi S, Tsuji O, Yamamoto T, Dunbar J. Diagnosis and management of idiopathic normal-pressure hydrocephalus: a prospective study in 151 patients. J Neurosurg. 2005 Jun;102(6):987-97. doi: 10.3171/jns.2005.102.6.0987. PMID 16028756
- [Background] Wikkelso C, Hellstrom P, Klinge PM, Tans JT; European iNPH Multicentre Study Group. The European iNPH Multicentre Study on the predictive values of resistance to CSF outflow and the CSF Tap Test in patients with idiopathic normal pressure hydrocephalus. J Neurol Neurosurg Psychiatry. 2013 May;84(5):562-8. doi: 10.1136/jnnp-2012-303314. Epub 2012 Dec 18. PMID 23250963
- [Background] Giannini G, Palandri G, Ferrari A, Oppi F, Milletti D, Albini-Riccioli L, Mantovani P, Magnoni S, Chiari L, Cortelli P, Cevoli S; BOLOGNA PRO-HYDRO Study Group. A prospective evaluation of clinical and instrumental features before and after ventriculo-peritoneal shunt in patients with idiopathic Normal pressure hydrocephalus: The Bologna PRO-Hydro study. Parkinsonism Relat Disord. 2019 Sep;66:117-124. doi: 10.1016/j.parkreldis.2019.07.021. Epub 2019 Jul 18. PMID 31358442
- [Background] Hebb AO, Cusimano MD. Idiopathic normal pressure hydrocephalus: a systematic review of diagnosis and outcome. Neurosurgery. 2001 Nov;49(5):1166-84; discussion 1184-6. doi: 10.1097/00006123-200111000-00028. PMID 11846911
- [Background] Mostile G, Fasano A, Zappia M. Parkinsonism in idiopathic normal pressure hydrocephalus: is it time for defining a clinical tetrad? Neurol Sci. 2022 Sep;43(9):5201-5205. doi: 10.1007/s10072-022-06119-3. Epub 2022 Jun 1. PMID 35648268
- [Background] Akiguchi I, Ishii M, Watanabe Y, Watanabe T, Kawasaki T, Yagi H, Shiino A, Shirakashi Y, Kawamoto Y. Shunt-responsive parkinsonism and reversible white matter lesions in patients with idiopathic NPH. J Neurol. 2008 Sep;255(9):1392-9. doi: 10.1007/s00415-008-0928-1. Epub 2008 Jun 27. PMID 18575921
- [Background] Todisco M, Zangaglia R, Minafra B, Pisano P, Trifiro G, Bossert I, Pozzi NG, Brumberg J, Ceravolo R, Isaias IU, Fasano A, Pacchetti C. Clinical Outcome and Striatal Dopaminergic Function After Shunt Surgery in Patients With Idiopathic Normal Pressure Hydrocephalus. Neurology. 2021 Jun 8;96(23):e2861-e2873. doi: 10.1212/WNL.0000000000012064. Epub 2021 Apr 23. PMID 33893195
- [Background] Nakayama T, Ouchi Y, Yoshikawa E, Sugihara G, Torizuka T, Tanaka K. Striatal D2 receptor availability after shunting in idiopathic normal pressure hydrocephalus. J Nucl Med. 2007 Dec;48(12):1981-6. doi: 10.2967/jnumed.107.045310. Epub 2007 Nov 15. PMID 18006609
- [Background] Ouchi Y, Nakayama T, Kanno T, Yoshikawa E, Shinke T, Torizuka T. In vivo presynaptic and postsynaptic striatal dopamine functions in idiopathic normal pressure hydrocephalus. J Cereb Blood Flow Metab. 2007 Apr;27(4):803-10. doi: 10.1038/sj.jcbfm.9600389. Epub 2006 Aug 16. PMID 16926840
- [Background] Curran T, Lang AE. Parkinsonian syndromes associated with hydrocephalus: case reports, a review of the literature, and pathophysiological hypotheses. Mov Disord. 1994 Sep;9(5):508-20. doi: 10.1002/mds.870090503. PMID 7990846
- [Background] Nakajima M, Yamada S, Miyajima M, Ishii K, Kuriyama N, Kazui H, Kanemoto H, Suehiro T, Yoshiyama K, Kameda M, Kajimoto Y, Mase M, Murai H, Kita D, Kimura T, Samejima N, Tokuda T, Kaijima M, Akiba C, Kawamura K, Atsuchi M, Hirata Y, Matsumae M, Sasaki M, Yamashita F, Aoki S, Irie R, Miyake H, Kato T, Mori E, Ishikawa M, Date I, Arai H; research committee of idiopathic normal pressure hydrocephalus. Guidelines for Management of Idiopathic Normal Pressure Hydrocephalus (Third Edition): Endorsed by the Japanese Society of Normal Pressure Hydrocephalus. Neurol Med Chir (Tokyo). 2021 Feb 15;61(2):63-97. doi: 10.2176/nmc.st.2020-0292. Epub 2021 Jan 15. PMID 33455998
- [Background] Krauss JK, Regel JP, Droste DW, Orszagh M, Borremans JJ, Vach W. Movement disorders in adult hydrocephalus. Mov Disord. 1997 Jan;12(1):53-60. doi: 10.1002/mds.870120110. PMID 8990054
- [Background] Molde K, Soderstrom L, Laurell K. Parkinsonian symptoms in normal pressure hydrocephalus: a population-based study. J Neurol. 2017 Oct;264(10):2141-2148. doi: 10.1007/s00415-017-8598-5. Epub 2017 Sep 6. PMID 28879446
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] Allali G, Annweiler C, Blumen HM, Callisaya ML, De Cock AM, Kressig RW, Srikanth V, Steinmetz JP, Verghese J, Beauchet O. Gait phenotype from mild cognitive impairment to moderate dementia: results from the GOOD initiative. Eur J Neurol. 2016 Mar;23(3):527-41. doi: 10.1111/ene.12882. Epub 2015 Dec 14. PMID 26662508
- [Background] Ishii M, Kawamata T, Akiguchi I, Yagi H, Watanabe Y, Watanabe T, Mashimo H. Parkinsonian Symptomatology May Correlate with CT Findings before and after Shunting in Idiopathic Normal Pressure Hydrocephalus. Parkinsons Dis. 2010 Mar 10;2010:201089. doi: 10.4061/2010/201089. PMID 20948890
- [Background] Kang K, Jeon JS, Kim T, Choi D, Ko PW, Hwang SK, Lee HW. Asymmetric and Upper Body Parkinsonism in Patients with Idiopathic Normal-Pressure Hydrocephalus. J Clin Neurol. 2016 Oct;12(4):452-459. doi: 10.3988/jcn.2016.12.4.452. Epub 2016 Jul 26. PMID 27486933
- [Background] Mostile G, Portaro G, Certo F, Luca A, Manna R, Terranova R, Altieri R, Nicoletti A, Barbagallo GMV, Zappia M. iNPH with parkinsonism: response to lumbar CSF drainage and ventriculoperitoneal shunting. J Neurol. 2021 Apr;268(4):1254-1265. doi: 10.1007/s00415-020-10267-x. Epub 2020 Oct 19. PMID 33078308
- [Background] Morishita T, Foote KD, Okun MS. INPH and Parkinson disease: differentiation by levodopa response. Nat Rev Neurol. 2010 Jan;6(1):52-6. doi: 10.1038/nrneurol.2009.195. PMID 20057498
- [Background] Youn J, Todisco M, Zappia M, Pacchetti C, Fasano A. Parkinsonism and cerebrospinal fluid disorders. J Neurol Sci. 2022 Feb 15;433:120019. doi: 10.1016/j.jns.2021.120019. Epub 2021 Oct 1. PMID 34674853
- [Background] Israelsson H, Allard P, Eklund A, Malm J. Symptoms of Depression are Common in Patients With Idiopathic Normal Pressure Hydrocephalus: The INPH-CRasH Study. Neurosurgery. 2016 Feb;78(2):161-8. doi: 10.1227/NEU.0000000000001093. PMID 26528670
- [Background] Bloom KK, Kraft WA. Paranoia--an unusual presentation of hydrocephalus. Am J Phys Med Rehabil. 1998 Mar-Apr;77(2):157-9. PMID 9558018
- [Background] Crowell RM, Tew JM Jr, Mark VH. Aggressive dementia associated with normal pressure hydrocephalus. Report of two unusual cases. Neurology. 1973 May;23(5):461-4. doi: 10.1212/wnl.23.5.461. No abstract available. PMID 4735461
- [Background] Yusim A, Anbarasan D, Bernstein C, Boksay I, Dulchin M, Lindenmayer JP, Saavedra-Velez C, Shapiro M, Sadock B. Normal pressure hydrocephalus presenting as Othello syndrome: case presentation and review of the literature. Am J Psychiatry. 2008 Sep;165(9):1119-25. doi: 10.1176/appi.ajp.2008.07111820. No abstract available. PMID 18765494
- [Background] Schneider U, Malmadier A, Dengler R, Sollmann WP, Emrich HM. Mood cycles associated with normal pressure hydrocephalus. Am J Psychiatry. 1996 Oct;153(10):1366-7. doi: 10.1176/ajp.153.10.1366. No abstract available. PMID 8831453
- [Background] Rosen H, Swigar ME. Depression and normal pressure hydrocephalus. A dilemma in neuropsychiatric differential diagnosis. J Nerv Ment Dis. 1976 Jul;163(1):35-40. doi: 10.1097/00005053-197607000-00005. PMID 932710
- [Background] Saito M, Nishio Y, Kanno S, Uchiyama M, Hayashi A, Takagi M, Kikuchi H, Yamasaki H, Shimomura T, Iizuka O, Mori E. Cognitive profile of idiopathic normal pressure hydrocephalus. Dement Geriatr Cogn Dis Extra. 2011 Jan;1(1):202-11. doi: 10.1159/000328924. Epub 2011 Jul 15. PMID 22163245
- [Background] Campos-Juanatey F, Gutierrez-Banos JL, Portillo-Martin JA, Zubillaga-Guerrero S. Assessment of the urodynamic diagnosis in patients with urinary incontinence associated with normal pressure hydrocephalus. Neurourol Urodyn. 2015 Jun;34(5):465-8. doi: 10.1002/nau.22600. Epub 2014 Apr 12. PMID 24729303
- [Background] Mc Ardle R, Galna B, Donaghy P, Thomas A, Rochester L. Do Alzheimer's and Lewy body disease have discrete pathological signatures of gait? Alzheimers Dement. 2019 Oct;15(10):1367-1377. doi: 10.1016/j.jalz.2019.06.4953. Epub 2019 Sep 20. PMID 31548122
- [Background] Agarwal S, Gilbert R. Progressive Supranuclear Palsy. 2023 Mar 27. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK526098/ PMID 30252354
- [Background] Kim SM, Kim DH, Yang Y, Ha SW, Han JH. Gait Patterns in Parkinson's Disease with or without Cognitive Impairment. Dement Neurocogn Disord. 2018 Jun;17(2):57-65. doi: 10.12779/dnd.2018.17.2.57. Epub 2018 Jul 24. PMID 30906393
- [Background] Fraser C, Stark SW. Gait disorder in older adults: is it NPH? Nurse Pract. 2011 Mar;36(3):14-20; quiz 20-1. doi: 10.1097/01.NPR.0000393969.13812.2e. PMID 21307803
- [Background] Williams MA, Nagel SJ, Luciano MG, Relkin N, Zwimpfer TJ, Katzen H, Holubkov R, Moghekar A, Wisoff JH, McKhann GM, Golomb J, Edwards RJ, Hamilton MG. The clinical spectrum of hydrocephalus in adults: report of the first 517 patients of the Adult Hydrocephalus Clinical Research Network registry. J Neurosurg. 2019 May 24;132(6):1773-1784. doi: 10.3171/2019.2.JNS183538. Print 2020 Jun 1. PMID 31125971
- [Background] Marmarou A, Bergsneider M, Relkin N, Klinge P, Black PM. Development of guidelines for idiopathic normal-pressure hydrocephalus: introduction. Neurosurgery. 2005 Sep;57(3 Suppl):S1-3; discussion ii-v. doi: 10.1227/01.neu.0000168188.25559.0e. PMID 16160424
- [Background] Williams MA, Malm J. Diagnosis and Treatment of Idiopathic Normal Pressure Hydrocephalus. Continuum (Minneap Minn). 2016 Apr;22(2 Dementia):579-99. doi: 10.1212/CON.0000000000000305. PMID 27042909
- [Background] Broggi M, Redaelli V, Tringali G, Restelli F, Romito L, Schiavolin S, Tagliavini F, Broggi G. Normal Pressure Hydrocephalus and Parkinsonism: Preliminary Data on Neurosurgical and Neurological Treatment. World Neurosurg. 2016 Jun;90:348-356. doi: 10.1016/j.wneu.2016.03.004. Epub 2016 Mar 10. PMID 26970480
- [Background] Knutsson E, Lying-Tunell U. Gait apraxia in normal-pressure hydrocephalus: patterns of movement and muscle activation. Neurology. 1985 Feb;35(2):155-60. doi: 10.1212/wnl.35.2.155. PMID 3969202
- [Background] Yoshino M, Yoshimi Y, Taniguchi M, Nakamura S, Ikeda T. Syndrome of inappropriate secretion of antidiuretic hormone associated with idiopathic normal pressure hydrocephalus. Intern Med. 1999 Mar;38(3):290-2. doi: 10.2169/internalmedicine.38.290. PMID 10337945
- [Background] Marmarou A, Black P, Bergsneider M, Klinge P, Relkin N; International NPH Consultant Group. Guidelines for management of idiopathic normal pressure hydrocephalus: progress to date. Acta Neurochir Suppl. 2005;95:237-40. doi: 10.1007/3-211-32318-x_48. PMID 16463856
- [Background] Isaacs AM, Williams MA, Hamilton MG. Current Update on Treatment Strategies for Idiopathic Normal Pressure Hydrocephalus. Curr Treat Options Neurol. 2019 Dec 3;21(12):65. doi: 10.1007/s11940-019-0604-z. PMID 31792620
- [Background] Pyykko OT, Helisalmi S, Koivisto AM, Molsa JA, Rummukainen J, Nerg O, Alafuzoff I, Savolainen S, Soininen H, Jaaskelainen JE, Rinne J, Leinonen V, Hiltunen M. APOE4 predicts amyloid-beta in cortical brain biopsy but not idiopathic normal pressure hydrocephalus. J Neurol Neurosurg Psychiatry. 2012 Nov;83(11):1119-24. doi: 10.1136/jnnp-2011-303849. Epub 2012 Sep 6. PMID 22955176
- [Background] Gudmundsson G, Kristjansdottir G, Cook E, Olafsson I. Association of ApoE genotype with clinical features and outcome in idiopathic normal pressure hydrocephalus (iNPH): a preliminary report. Acta Neurochir (Wien). 2009 Nov;151(11):1511-2. doi: 10.1007/s00701-009-0429-8. Epub 2009 Jun 24. PMID 19551336
- [Background] Cusimano MD, Rewilak D, Stuss DT, Barrera-Martinez JC, Salehi F, Freedman M. Normal-pressure hydrocephalus: is there a genetic predisposition? Can J Neurol Sci. 2011 Mar;38(2):274-81. doi: 10.1017/s031716710001146x. PMID 21320833
- [Background] Korhonen VE, Helisalmi S, Jokinen A, Jokinen I, Lehtola JM, Oinas M, Lonnrot K, Avellan C, Kotkansalo A, Frantzen J, Rinne J, Ronkainen A, Kauppinen M, Junkkari A, Hiltunen M, Soininen H, Kurki M, Jaaskelainen JE, Koivisto AM, Sato H, Kato T, Remes AM, Eide PK, Leinonen V. Copy number loss in SFMBT1 is common among Finnish and Norwegian patients with iNPH. Neurol Genet. 2018 Dec 3;4(6):e291. doi: 10.1212/NXG.0000000000000291. eCollection 2018 Dec. PMID 30584596
- [Background] Sato H, Takahashi Y, Kimihira L, Iseki C, Kato H, Suzuki Y, Igari R, Sato H, Koyama S, Arawaka S, Kawanami T, Miyajima M, Samejima N, Sato S, Kameda M, Yamada S, Kita D, Kaijima M, Date I, Sonoda Y, Kayama T, Kuwana N, Arai H, Kato T. A Segmental Copy Number Loss of the SFMBT1 Gene Is a Genetic Risk for Shunt-Responsive, Idiopathic Normal Pressure Hydrocephalus (iNPH): A Case-Control Study. PLoS One. 2016 Nov 18;11(11):e0166615. doi: 10.1371/journal.pone.0166615. eCollection 2016. PMID 27861535
- [Background] Zhang J, Bonasio R, Strino F, Kluger Y, Holloway JK, Modzelewski AJ, Cohen PE, Reinberg D. SFMBT1 functions with LSD1 to regulate expression of canonical histone genes and chromatin-related factors. Genes Dev. 2013 Apr 1;27(7):749-66. doi: 10.1101/gad.210963.112. PMID 23592795
- [Background] Kato T, Sato H, Emi M, Seino T, Arawaka S, Iseki C, Takahashi Y, Wada M, Kawanami T. Segmental copy number loss of SFMBT1 gene in elderly individuals with ventriculomegaly: a community-based study. Intern Med. 2011;50(4):297-303. doi: 10.2169/internalmedicine.50.4505. Epub 2011 Feb 15. PMID 21325761
- [Background] Morimoto Y, Yoshida S, Kinoshita A, Satoh C, Mishima H, Yamaguchi N, Matsuda K, Sakaguchi M, Tanaka T, Komohara Y, Imamura A, Ozawa H, Nakashima M, Kurotaki N, Kishino T, Yoshiura KI, Ono S. Nonsense mutation in CFAP43 causes normal-pressure hydrocephalus with ciliary abnormalities. Neurology. 2019 May 14;92(20):e2364-e2374. doi: 10.1212/WNL.0000000000007505. Epub 2019 Apr 19. PMID 31004071
- [Background] Duriez B, Duquesnoy P, Escudier E, Bridoux AM, Escalier D, Rayet I, Marcos E, Vojtek AM, Bercher JF, Amselem S. A common variant in combination with a nonsense mutation in a member of the thioredoxin family causes primary ciliary dyskinesia. Proc Natl Acad Sci U S A. 2007 Feb 27;104(9):3336-41. doi: 10.1073/pnas.0611405104. Epub 2007 Feb 20. PMID 17360648
- [Background] Liouta E, Liakos F, Koutsarnakis C, Katsaros V, Stranjalis G. Novel case of familial normal pressure hydrocephalus. Psychiatry Clin Neurosci. 2014 Jul;68(7):583-4. doi: 10.1111/pcn.12176. Epub 2014 Apr 14. No abstract available. PMID 24612122
- [Background] Takahashi Y, Kawanami T, Nagasawa H, Iseki C, Hanyu H, Kato T. Familial normal pressure hydrocephalus (NPH) with an autosomal-dominant inheritance: a novel subgroup of NPH. J Neurol Sci. 2011 Sep 15;308(1-2):149-51. doi: 10.1016/j.jns.2011.06.018. Epub 2011 Jun 24. PMID 21704338
- [Background] Zhang J, Carr CW, Rigamonti D, Badr A. Genome-wide linkage scan maps ETINPH gene to chromosome 19q12-13.31. Hum Hered. 2010;69(4):262-7. doi: 10.1159/000288711. Epub 2010 Mar 31. PMID 20357477
- [Background] Zhang J, Williams MA, Rigamonti D. Heritable essential tremor-idiopathic normal pressure hydrocephalus (ETINPH). Am J Med Genet A. 2008 Feb 15;146A(4):433-9. doi: 10.1002/ajmg.a.31958. PMID 18203159
- [Background] Huovinen J, Kastinen S, Komulainen S, Oinas M, Avellan C, Frantzen J, Rinne J, Ronkainen A, Kauppinen M, Lonnrot K, Perola M, Pyykko OT, Koivisto AM, Remes AM, Soininen H, Hiltunen M, Helisalmi S, Kurki M, Jaaskelainen JE, Leinonen V. Familial idiopathic normal pressure hydrocephalus. J Neurol Sci. 2016 Sep 15;368:11-8. doi: 10.1016/j.jns.2016.06.052. Epub 2016 Jun 25. PMID 27538594
- [Background] McGirr A, Cusimano MD. Familial aggregation of idiopathic normal pressure hydrocephalus: novel familial case and a family study of the NPH triad in an iNPH patient cohort. J Neurol Sci. 2012 Oct 15;321(1-2):82-8. doi: 10.1016/j.jns.2012.07.062. Epub 2012 Aug 23. PMID 22921954
- [Background] Oliveira MF, Nacif SR, Castellano O, Sousa UO, Rotta JM, Pinto FC. Improvement of Central Sleep Apneas Following Ventricular Shunt for Normal Pressure Hydrocephalus. J Neuropsychiatry Clin Neurosci. 2015 Summer;27(3):e206-8. doi: 10.1176/appi.neuropsych.14120375. No abstract available. PMID 26222970
- [Background] Kuchiwaki H, Kageyama N, Hirai N, Takada S, Inao S, Terashima M, Sugiura M. [A biological rhythm in a patient with normal pressure hydrocephalus--comparative studies in pre- and postoperative patients by a polygraphy]. No To Shinkei. 1984 Sep;36(9):911-6. Japanese. PMID 6508959
- [Background] Roman GC, Jackson RE, Fung SH, Zhang YJ, Verma AK. Sleep-Disordered Breathing and Idiopathic Normal-Pressure Hydrocephalus: Recent Pathophysiological Advances. Curr Neurol Neurosci Rep. 2019 May 29;19(7):39. doi: 10.1007/s11910-019-0952-9. PMID 31144048
- [Background] Ooms S, Ju YE. Treatment of Sleep Disorders in Dementia. Curr Treat Options Neurol. 2016 Sep;18(9):40. doi: 10.1007/s11940-016-0424-3. PMID 27476067
- [Background] Lee MJ, Chang CP, Lee YH, Wu YC, Tseng HW, Tung YY, Wu MT, Chen YH, Kuo LT, Stephenson D, Hung SI, Wu JY, Chang C, Chen YT, Chern Y. Longitudinal evaluation of an N-ethyl-N-nitrosourea-created murine model with normal pressure hydrocephalus. PLoS One. 2009 Nov 17;4(11):e7868. doi: 10.1371/journal.pone.0007868. PMID 19924295
- [Background] Sharma S, Goyal MK, Sharma K, Modi M, Sharma M, Khandelwal N, Prabhakar S, Sharma N, R S, Gairolla J, Jain A, Lal V. Cytokines do play a role in pathogenesis of tuberculous meningitis: A prospective study from a tertiary care center in India. J Neurol Sci. 2017 Aug 15;379:131-136. doi: 10.1016/j.jns.2017.06.001. Epub 2017 Jun 3. PMID 28716226
- [Background] Eide PK, Sorteberg W. Outcome of Surgery for Idiopathic Normal Pressure Hydrocephalus: Role of Preoperative Static and Pulsatile Intracranial Pressure. World Neurosurg. 2016 Feb;86:186-193.e1. doi: 10.1016/j.wneu.2015.09.067. Epub 2015 Sep 30. PMID 26428326
- [Background] Koivisto AM, Alafuzoff I, Savolainen S, Sutela A, Rummukainen J, Kurki M, Jaaskelainen JE, Soininen H, Rinne J, Leinonen V; Kuopio NPH Registry (www.uef.finph). Poor cognitive outcome in shunt-responsive idiopathic normal pressure hydrocephalus. Neurosurgery. 2013 Jan;72(1):1-8;discussion 8. doi: 10.1227/NEU.0b013e31827414b3. PMID 23037817
- [Background] Hamilton R, Patel S, Lee EB, Jackson EM, Lopinto J, Arnold SE, Clark CM, Basil A, Shaw LM, Xie SX, Grady MS, Trojanowski JQ. Lack of shunt response in suspected idiopathic normal pressure hydrocephalus with Alzheimer disease pathology. Ann Neurol. 2010 Oct;68(4):535-40. doi: 10.1002/ana.22015. PMID 20687117
- [Background] Thaker AA, Weinberg BD, Dillon WP, Hess CP, Cabral HJ, Fleischman DA, Leurgans SE, Bennett DA, Hyman BT, Albert MS, Killiany RJ, Fischl B, Dale AM, Desikan RS. Entorhinal Cortex: Antemortem Cortical Thickness and Postmortem Neurofibrillary Tangles and Amyloid Pathology. AJNR Am J Neuroradiol. 2017 May;38(5):961-965. doi: 10.3174/ajnr.A5133. Epub 2017 Mar 9. PMID 28279988
- [Background] Hyman BT, Van Hoesen GW, Damasio AR, Barnes CL. Alzheimer's disease: cell-specific pathology isolates the hippocampal formation. Science. 1984 Sep 14;225(4667):1168-70. doi: 10.1126/science.6474172.
- [Background] Rasmussen MK, Mestre H, Nedergaard M. The glymphatic pathway in neurological disorders. Lancet Neurol. 2018 Nov;17(11):1016-1024. doi: 10.1016/S1474-4422(18)30318-1. PMID 30353860
- [Background] Shook BA, Lennington JB, Acabchuk RL, Halling M, Sun Y, Peters J, Wu Q, Mahajan A, Fellows DW, Conover JC. Ventriculomegaly associated with ependymal gliosis and declines in barrier integrity in the aging human and mouse brain. Aging Cell. 2014 Apr;13(2):340-50. doi: 10.1111/acel.12184. Epub 2013 Dec 17. PMID 24341850
- [Background] Yamada S, Ishikawa M, Ito H, Yamamoto K, Yamaguchi M, Oshima M, Nozaki K. Cerebrospinal fluid dynamics in idiopathic normal pressure hydrocephalus on four-dimensional flow imaging. Eur Radiol. 2020 Aug;30(8):4454-4465. doi: 10.1007/s00330-020-06825-6. Epub 2020 Apr 3. PMID 32246220
- [Background] Eide PK, Lashkarivand A, Hagen-Kersten AA, Gjertsen O, Nedregaard B, Sletteberg R, Lovland G, Vatnehol SAS, Pripp AH, Valnes LM, Ringstad G. Intrathecal Contrast-Enhanced Magnetic Resonance Imaging of Cerebrospinal Fluid Dynamics and Glymphatic Enhancement in Idiopathic Normal Pressure Hydrocephalus. Front Neurol. 2022 Apr 6;13:857328. doi: 10.3389/fneur.2022.857328. eCollection 2022. PMID 35463139
- [Background] Eide PK, Vatnehol SAS, Emblem KE, Ringstad G. Magnetic resonance imaging provides evidence of glymphatic drainage from human brain to cervical lymph nodes. Sci Rep. 2018 May 8;8(1):7194. doi: 10.1038/s41598-018-25666-4. PMID 29740121
- [Background] Louveau A, Plog BA, Antila S, Alitalo K, Nedergaard M, Kipnis J. Understanding the functions and relationships of the glymphatic system and meningeal lymphatics. J Clin Invest. 2017 Sep 1;127(9):3210-3219. doi: 10.1172/JCI90603. Epub 2017 Sep 1. PMID 28862640
- [Background] Iliff JJ, Wang M, Zeppenfeld DM, Venkataraman A, Plog BA, Liao Y, Deane R, Nedergaard M. Cerebral arterial pulsation drives paravascular CSF-interstitial fluid exchange in the murine brain. J Neurosci. 2013 Nov 13;33(46):18190-9. doi: 10.1523/JNEUROSCI.1592-13.2013. PMID 24227727
- [Background] Roher AE, Esh C, Kokjohn TA, Kalback W, Luehrs DC, Seward JD, Sue LI, Beach TG. Circle of willis atherosclerosis is a risk factor for sporadic Alzheimer's disease. Arterioscler Thromb Vasc Biol. 2003 Nov 1;23(11):2055-62. doi: 10.1161/01.ATV.0000095973.42032.44. Epub 2003 Sep 25. PMID 14512367
- [Background] Eide PK, Sorteberg W. Diagnostic intracranial pressure monitoring and surgical management in idiopathic normal pressure hydrocephalus: a 6-year review of 214 patients. Neurosurgery. 2010 Jan;66(1):80-91. doi: 10.1227/01.NEU.0000363408.69856.B8. PMID 20023540
- [Background] Greitz D. Radiological assessment of hydrocephalus: new theories and implications for therapy. Neurosurg Rev. 2004 Jul;27(3):145-65; discussion 166-7. doi: 10.1007/s10143-004-0326-9. Epub 2004 May 26. PMID 15164255
- [Background] Picascia M, Zangaglia R, Bernini S, Minafra B, Sinforiani E, Pacchetti C. A review of cognitive impairment and differential diagnosis in idiopathic normal pressure hydrocephalus. Funct Neurol. 2015 Oct-Dec;30(4):217-28. doi: 10.11138/fneur/2015.30.4.217. PMID 26727700
- [Background] Andersson KE. Mechanisms of Disease: central nervous system involvement in overactive bladder syndrome. Nat Clin Pract Urol. 2004 Dec;1(2):103-8. doi: 10.1038/ncpuro0021. PMID 16474523
- [Background] Momjian S, Owler BK, Czosnyka Z, Czosnyka M, Pena A, Pickard JD. Pattern of white matter regional cerebral blood flow and autoregulation in normal pressure hydrocephalus. Brain. 2004 May;127(Pt 5):965-72. doi: 10.1093/brain/awh131. Epub 2004 Mar 19. PMID 15033897
- [Background] Owler BK, Pickard JD. Normal pressure hydrocephalus and cerebral blood flow: a review. Acta Neurol Scand. 2001 Dec;104(6):325-42. doi: 10.1034/j.1600-0404.2001.00092.x. PMID 11903086
- [Background] Owler BK, Momjian S, Czosnyka Z, Czosnyka M, Pena A, Harris NG, Smielewski P, Fryer T, Donovan T, Coles J, Carpenter A, Pickard JD. Normal pressure hydrocephalus and cerebral blood flow: a PET study of baseline values. J Cereb Blood Flow Metab. 2004 Jan;24(1):17-23. doi: 10.1097/01.WCB.0000093326.88757.49. PMID 14688613
- [Background] Ziegelitz D, Starck G, Kristiansen D, Jakobsson M, Hultenmo M, Mikkelsen IK, Hellstrom P, Tullberg M, Wikkelso C. Cerebral perfusion measured by dynamic susceptibility contrast MRI is reduced in patients with idiopathic normal pressure hydrocephalus. J Magn Reson Imaging. 2014 Jun;39(6):1533-42. doi: 10.1002/jmri.24292. Epub 2013 Sep 4. PMID 24006249
- [Background] Virhammar J, Laurell K, Ahlgren A, Larsson EM. Arterial Spin-Labeling Perfusion MR Imaging Demonstrates Regional CBF Decrease in Idiopathic Normal Pressure Hydrocephalus. AJNR Am J Neuroradiol. 2017 Nov;38(11):2081-2088. doi: 10.3174/ajnr.A5347. Epub 2017 Aug 31. PMID 28860216
- [Background] Krauss JK, Regel JP, Vach W, Orszagh M, Jungling FD, Bohus M, Droste DW. White matter lesions in patients with idiopathic normal pressure hydrocephalus and in an age-matched control group: a comparative study. Neurosurgery. 1997 Mar;40(3):491-5; discussion 495-6. doi: 10.1097/00006123-199703000-00011. PMID 9055287
- [Background] Eide PK, Pripp AH. Increased prevalence of cardiovascular disease in idiopathic normal pressure hydrocephalus patients compared to a population-based cohort from the HUNT3 survey. Fluids Barriers CNS. 2014 Aug 19;11:19. doi: 10.1186/2045-8118-11-19. eCollection 2014. PMID 25180074
- [Background] Jacobs L. Diabetes mellitus in normal pressure hydrocephalus. J Neurol Neurosurg Psychiatry. 1977 Apr;40(4):331-5. doi: 10.1136/jnnp.40.4.331. PMID 874510
- [Background] Krauss JK, Regel JP, Vach W, Droste DW, Borremans JJ, Mergner T. Vascular risk factors and arteriosclerotic disease in idiopathic normal-pressure hydrocephalus of the elderly. Stroke. 1996 Jan;27(1):24-9. doi: 10.1161/01.str.27.1.24. PMID 8553398
- [Background] Hickman TT, Shuman ME, Johnson TA, Yang F, Rice RR, Rice IM, Chung EH, Wiemann R, Tinl M, Iracheta C, Chen G, Flynn P, Mondello MB, Thompson J, Meadows ME, Carroll RS, Yang HW, Xing H, Pilgrim D, Chiocca EA, Dunn IF, Golby AJ, Johnson MD. Association between shunt-responsive idiopathic normal pressure hydrocephalus and alcohol. J Neurosurg. 2017 Aug;127(2):240-248. doi: 10.3171/2016.6.JNS16496. Epub 2016 Sep 30. PMID 27689463
- [Background] Stephensen H, Andersson N, Eklund A, Malm J, Tisell M, Wikkelso C. Objective B wave analysis in 55 patients with non-communicating and communicating hydrocephalus. J Neurol Neurosurg Psychiatry. 2005 Jul;76(7):965-70. doi: 10.1136/jnnp.2004.039834. PMID 15965203
- [Background] Marmarou A, Young HF, Aygok GA. Estimated incidence of normal pressure hydrocephalus and shunt outcome in patients residing in assisted-living and extended-care facilities. Neurosurg Focus. 2007 Apr 15;22(4):E1. doi: 10.3171/foc.2007.22.4.2. PMID 17613187
- [Background] Brean A, Fredo HL, Sollid S, Muller T, Sundstrom T, Eide PK. Five-year incidence of surgery for idiopathic normal pressure hydrocephalus in Norway. Acta Neurol Scand. 2009 Nov;120(5):314-6. doi: 10.1111/j.1600-0404.2009.01250.x. PMID 19832773
- [Background] Tisell M, Hoglund M, Wikkelso C. National and regional incidence of surgery for adult hydrocephalus in Sweden. Acta Neurol Scand. 2005 Aug;112(2):72-5. doi: 10.1111/j.1600-0404.2005.00451.x. PMID 16008530
- [Background] Vanneste J, Augustijn P, Dirven C, Tan WF, Goedhart ZD. Shunting normal-pressure hydrocephalus: do the benefits outweigh the risks? A multicenter study and literature review. Neurology. 1992 Jan;42(1):54-9. doi: 10.1212/wnl.42.1.54. PMID 1734324
- [Background] Kuriyama N, Miyajima M, Nakajima M, Kurosawa M, Fukushima W, Watanabe Y, Ozaki E, Hirota Y, Tamakoshi A, Mori E, Kato T, Tokuda T, Urae A, Arai H. Nationwide hospital-based survey of idiopathic normal pressure hydrocephalus in Japan: Epidemiological and clinical characteristics. Brain Behav. 2017 Jan 27;7(3):e00635. doi: 10.1002/brb3.635. eCollection 2017 Mar. PMID 28293475
- [Background] Tanaka N, Yamaguchi S, Ishikawa H, Ishii H, Meguro K. Prevalence of possible idiopathic normal-pressure hydrocephalus in Japan: the Osaki-Tajiri project. Neuroepidemiology. 2009;32(3):171-5. doi: 10.1159/000186501. Epub 2008 Dec 19. PMID 19096225
- [Background] Andersson J, Rosell M, Kockum K, Lilja-Lund O, Soderstrom L, Laurell K. Prevalence of idiopathic normal pressure hydrocephalus: A prospective, population-based study. PLoS One. 2019 May 29;14(5):e0217705. doi: 10.1371/journal.pone.0217705. eCollection 2019. PMID 31141553
- [Background] Yang HW, Lee S, Yang D, Dai H, Zhang Y, Han L, Zhao S, Zhang S, Ma Y, Johnson MF, Rattray AK, Johnson TA, Wang G, Zheng S, Carroll RS, Park PJ, Johnson MD. Deletions in CWH43 cause idiopathic normal pressure hydrocephalus. EMBO Mol Med. 2021 Mar 5;13(3):e13249. doi: 10.15252/emmm.202013249. Epub 2021 Jan 18. PMID 33459505
- [Background] Kiefer M, Unterberg A. The differential diagnosis and treatment of normal-pressure hydrocephalus. Dtsch Arztebl Int. 2012 Jan;109(1-2):15-25; quiz 26. doi: 10.3238/arztebl.2012.0015. Epub 2012 Jan 9. PMID 22282714
- [Background] Martin-Laez R, Caballero-Arzapalo H, Valle-San Roman N, Lopez-Menendez LA, Arango-Lasprilla JC, Vazquez-Barquero A. Incidence of Idiopathic Normal-Pressure Hydrocephalus in Northern Spain. World Neurosurg. 2016 Mar;87:298-310. doi: 10.1016/j.wneu.2015.10.069. Epub 2015 Nov 5. PMID 26548835
- [Background] Zaccaria V, Bacigalupo I, Gervasi G, Canevelli M, Corbo M, Vanacore N, Lacorte E. A systematic review on the epidemiology of normal pressure hydrocephalus. Acta Neurol Scand. 2020 Feb;141(2):101-114. doi: 10.1111/ane.13182. Epub 2019 Nov 21. PMID 31622497
- [Background] Jaraj D, Rabiei K, Marlow T, Jensen C, Skoog I, Wikkelso C. Prevalence of idiopathic normal-pressure hydrocephalus. Neurology. 2014 Apr 22;82(16):1449-54. doi: 10.1212/WNL.0000000000000342. Epub 2014 Mar 28. PMID 24682964
- [Background] Brean A, Eide PK. Prevalence of probable idiopathic normal pressure hydrocephalus in a Norwegian population. Acta Neurol Scand. 2008 Jul;118(1):48-53. doi: 10.1111/j.1600-0404.2007.00982.x. Epub 2008 Jan 16. PMID 18205881
- [Background] Reeves BC, Karimy JK, Kundishora AJ, Mestre H, Cerci HM, Matouk C, Alper SL, Lundgaard I, Nedergaard M, Kahle KT. Glymphatic System Impairment in Alzheimer's Disease and Idiopathic Normal Pressure Hydrocephalus. Trends Mol Med. 2020 Mar;26(3):285-295. doi: 10.1016/j.molmed.2019.11.008. Epub 2020 Jan 18. PMID 31959516
- [Background] Ojemann RG, Fisher CM, Adams RD, Sweet WH, New PF. Further experience with the syndrome of "normal" pressure hydrocephalus. J Neurosurg. 1969 Sep;31(3):279-94. doi: 10.3171/jns.1969.31.3.0279. No abstract available. PMID 5811831
- [Background] Relkin N, Marmarou A, Klinge P, Bergsneider M, Black PM. Diagnosing idiopathic normal-pressure hydrocephalus. Neurosurgery. 2005 Sep;57(3 Suppl):S4-16; discussion ii-v. doi: 10.1227/01.neu.0000168185.29659.c5. PMID 16160425
- [Background] Mori E, Ishikawa M, Kato T, Kazui H, Miyake H, Miyajima M, Nakajima M, Hashimoto M, Kuriyama N, Tokuda T, Ishii K, Kaijima M, Hirata Y, Saito M, Arai H; Japanese Society of Normal Pressure Hydrocephalus. Guidelines for management of idiopathic normal pressure hydrocephalus: second edition. Neurol Med Chir (Tokyo). 2012;52(11):775-809. doi: 10.2176/nmc.52.775. PMID 23183074
- [Background] Bech-Azeddine R, Waldemar G, Knudsen GM, Hogh P, Bruhn P, Wildschiodtz G, Gjerris F, Paulson OB, Juhler M. Idiopathic normal-pressure hydrocephalus: evaluation and findings in a multidisciplinary memory clinic. Eur J Neurol. 2001 Nov;8(6):601-11. doi: 10.1046/j.1468-1331.2001.00291.x. PMID 11784345
- [Background] Ding Y, Zhang T, Wu G, McBride DW, Xu N, Klebe DW, Zhang Y, Li Q, Tang J, Zhang JH. Astrogliosis inhibition attenuates hydrocephalus by increasing cerebrospinal fluid reabsorption through the glymphatic system after germinal matrix hemorrhage. Exp Neurol. 2019 Oct;320:113003. doi: 10.1016/j.expneurol.2019.113003. Epub 2019 Jun 28. PMID 31260658
- [Background] Gavrilov GV, Stanishevskiy AV, Gaydar BV, Paramonova NM, Gaykova ON, Svistov DV. [Pathological changes in human brain biopsies from patients with idiopathic normal pressure hydrocephalus]. Zh Nevrol Psikhiatr Im S S Korsakova. 2019;119(3):50-54. doi: 10.17116/jnevro201911903150. Russian. PMID 31089095
- [Background] Golomb J, Wisoff J, Miller DC, Boksay I, Kluger A, Weiner H, Salton J, Graves W. Alzheimer's disease comorbidity in normal pressure hydrocephalus: prevalence and shunt response. J Neurol Neurosurg Psychiatry. 2000 Jun;68(6):778-81. doi: 10.1136/jnnp.68.6.778. PMID 10811706
- [Background] Savolainen S, Paljarvi L, Vapalahti M. Prevalence of Alzheimer's disease in patients investigated for presumed normal pressure hydrocephalus: a clinical and neuropathological study. Acta Neurochir (Wien). 1999;141(8):849-53. doi: 10.1007/s007010050386. PMID 10536721
- [Background] Leinonen V, Koivisto AM, Savolainen S, Rummukainen J, Tamminen JN, Tillgren T, Vainikka S, Pyykko OT, Molsa J, Fraunberg M, Pirttila T, Jaaskelainen JE, Soininen H, Rinne J, Alafuzoff I. Amyloid and tau proteins in cortical brain biopsy and Alzheimer's disease. Ann Neurol. 2010 Oct;68(4):446-53. doi: 10.1002/ana.22100. PMID 20976765
- [Background] Pomeraniec IJ, Bond AE, Lopes MB, Jane JA Sr. Concurrent Alzheimer's pathology in patients with clinical normal pressure hydrocephalus: correlation of high-volume lumbar puncture results, cortical brain biopsies, and outcomes. J Neurosurg. 2016 Feb;124(2):382-8. doi: 10.3171/2015.2.JNS142318. Epub 2015 Sep 4. PMID 26339853
- [Background] McGirt MJ, Woodworth G, Coon AL, Thomas G, Williams MA, Rigamonti D. Diagnosis, treatment, and analysis of long-term outcomes in idiopathic normal-pressure hydrocephalus. Neurosurgery. 2005 Oct;57(4):699-705; discussion 699-705. doi: 10.1093/neurosurgery/57.4.699. PMID 16239882
- [Background] Adams RD, Fisher CM, Hakim S, Ojemann RG, Sweet WH. SYMPTOMATIC OCCULT HYDROCEPHALUS WITH "NORMAL" CEREBROSPINAL-FLUID PRESSURE. A TREATABLE SYNDROME. N Engl J Med. 1965 Jul 15;273:117-26. doi: 10.1056/NEJM196507152730301. No abstract available. PMID 14303656
- [Background] Andersson J, Rosell M, Kockum K, Soderstrom L, Laurell K. Challenges in diagnosing normal pressure hydrocephalus: Evaluation of the diagnostic guidelines. eNeurologicalSci. 2017 Apr 11;7:27-31. doi: 10.1016/j.ensci.2017.04.002. eCollection 2017 Jun. PMID 29302622
- [Background] Yokota H, Vijayasarathi A, Cekic M, Hirata Y, Linetsky M, Ho M, Kim W, Salamon N. Diagnostic Performance of Glymphatic System Evaluation Using Diffusion Tensor Imaging in Idiopathic Normal Pressure Hydrocephalus and Mimickers. Curr Gerontol Geriatr Res. 2019 Jun 20;2019:5675014. doi: 10.1155/2019/5675014. eCollection 2019. PMID 31320896
- [Background] Kikuta J, Kamagata K, Taoka T, Takabayashi K, Uchida W, Saito Y, Andica C, Wada A, Kawamura K, Akiba C, Nakajima M, Miyajima M, Naganawa S, Aoki S. Water Diffusivity Changes Along the Perivascular Space After Lumboperitoneal Shunt Surgery in Idiopathic Normal Pressure Hydrocephalus. Front Neurol. 2022 Feb 28;13:843883. doi: 10.3389/fneur.2022.843883. eCollection 2022. PMID 35295837
- [Background] Bae YJ, Choi BS, Kim JM, Choi JH, Cho SJ, Kim JH. Altered glymphatic system in idiopathic normal pressure hydrocephalus. Parkinsonism Relat Disord. 2021 Jan;82:56-60. doi: 10.1016/j.parkreldis.2020.11.009. Epub 2020 Nov 20. PMID 33248394
- [Background] Carotenuto A, Cacciaguerra L, Pagani E, Preziosa P, Filippi M, Rocca MA. Glymphatic system impairment in multiple sclerosis: relation with brain damage and disability. Brain. 2022 Aug 27;145(8):2785-2795. doi: 10.1093/brain/awab454. PMID 34919648
- [Background] Cacciaguerra L, Carotenuto A, Pagani E, Mistri D, Radaelli M, Martinelli V, Filippi M, Rocca MA. Magnetic Resonance Imaging Evaluation of Perivascular Space Abnormalities in Neuromyelitis Optica. Ann Neurol. 2022 Aug;92(2):173-183. doi: 10.1002/ana.26419. Epub 2022 Jun 11. PMID 35596582
- [Background] Lee HJ, Lee DA, Shin KJ, Park KM. Glymphatic system dysfunction in obstructive sleep apnea evidenced by DTI-ALPS. Sleep Med. 2022 Jan;89:176-181. doi: 10.1016/j.sleep.2021.12.013. Epub 2021 Dec 28. PMID 35030357
- [Background] McKnight CD, Trujillo P, Lopez AM, Petersen K, Considine C, Lin YC, Yan Y, Kang H, Donahue MJ, Claassen DO. Diffusion along perivascular spaces reveals evidence supportive of glymphatic function impairment in Parkinson disease. Parkinsonism Relat Disord. 2021 Aug;89:98-104. doi: 10.1016/j.parkreldis.2021.06.004. Epub 2021 Jun 10. PMID 34271425
- [Background] Chen HL, Chen PC, Lu CH, Tsai NW, Yu CC, Chou KH, Lai YR, Taoka T, Lin WC. Associations among Cognitive Functions, Plasma DNA, and Diffusion Tensor Image along the Perivascular Space (DTI-ALPS) in Patients with Parkinson's Disease. Oxid Med Cell Longev. 2021 Feb 16;2021:4034509. doi: 10.1155/2021/4034509. eCollection 2021. PMID 33680283
- [Background] Siow TY, Toh CH, Hsu JL, Liu GH, Lee SH, Chen NH, Fu CJ, Castillo M, Fang JT. Association of Sleep, Neuropsychological Performance, and Gray Matter Volume With Glymphatic Function in Community-Dwelling Older Adults. Neurology. 2022 Feb 22;98(8):e829-e838. doi: 10.1212/WNL.0000000000013215. Epub 2021 Dec 14. PMID 34906982
- [Background] Taoka T, Fukusumi A, Miyasaka T, Kawai H, Nakane T, Kichikawa K, Naganawa S. Structure of the Medullary Veins of the Cerebral Hemisphere and Related Disorders. Radiographics. 2017 Jan-Feb;37(1):281-297. doi: 10.1148/rg.2017160061. PMID 28076020
- [Background] Komlosh ME, Benjamini D, Williamson NW, Horkay F, Hutchinson EB, Basser PJ. A novel MRI phantom to study interstitial fluid transport in the glymphatic system. Magn Reson Imaging. 2019 Feb;56:181-186. doi: 10.1016/j.mri.2018.10.007. Epub 2018 Oct 19. PMID 30343124
- [Background] Demiral SB, Tomasi D, Sarlls J, Lee H, Wiers CE, Zehra A, Srivastava T, Ke K, Shokri-Kojori E, Freeman CR, Lindgren E, Ramirez V, Miller G, Bandettini P, Horovitz S, Wang GJ, Benveniste H, Volkow ND. Apparent diffusion coefficient changes in human brain during sleep - Does it inform on the existence of a glymphatic system? Neuroimage. 2019 Jan 15;185:263-273. doi: 10.1016/j.neuroimage.2018.10.043. Epub 2018 Oct 17. PMID 30342236
- [Background] Thomas C, Sadeghi N, Nayak A, Trefler A, Sarlls J, Baker CI, Pierpaoli C. Impact of time-of-day on diffusivity measures of brain tissue derived from diffusion tensor imaging. Neuroimage. 2018 Jun;173:25-34. doi: 10.1016/j.neuroimage.2018.02.026. Epub 2018 Feb 16. PMID 29458189
- [Background] Harrison IF, Siow B, Akilo AB, Evans PG, Ismail O, Ohene Y, Nahavandi P, Thomas DL, Lythgoe MF, Wells JA. Non-invasive imaging of CSF-mediated brain clearance pathways via assessment of perivascular fluid movement with diffusion tensor MRI. Elife. 2018 Jul 31;7:e34028. doi: 10.7554/eLife.34028. PMID 30063207
- [Background] Chianca V, Albano D, Messina C, Cinnante CM, Triulzi FM, Sardanelli F, Sconfienza LM. Diffusion tensor imaging in the musculoskeletal and peripheral nerve systems: from experimental to clinical applications. Eur Radiol Exp. 2017;1(1):12. doi: 10.1186/s41747-017-0018-1. Epub 2017 Sep 30. PMID 29708174
- [Background] Tae WS, Ham BJ, Pyun SB, Kang SH, Kim BJ. Current Clinical Applications of Diffusion-Tensor Imaging in Neurological Disorders. J Clin Neurol. 2018 Apr;14(2):129-140. doi: 10.3988/jcn.2018.14.2.129. Epub 2018 Feb 28. PMID 29504292
- [Background] Taoka T, Masutani Y, Kawai H, Nakane T, Matsuoka K, Yasuno F, Kishimoto T, Naganawa S. Evaluation of glymphatic system activity with the diffusion MR technique: diffusion tensor image analysis along the perivascular space (DTI-ALPS) in Alzheimer's disease cases. Jpn J Radiol. 2017 Apr;35(4):172-178. doi: 10.1007/s11604-017-0617-z. Epub 2017 Feb 14. PMID 28197821
- [Background] Bechet NB, Kylkilahti TM, Mattsson B, Petrasova M, Shanbhag NC, Lundgaard I. Light sheet fluorescence microscopy of optically cleared brains for studying the glymphatic system. J Cereb Blood Flow Metab. 2020 Oct;40(10):1975-1986. doi: 10.1177/0271678X20924954. Epub 2020 Jun 11. PMID 32525440
- [Background] Iliff JJ, Lee H, Yu M, Feng T, Logan J, Nedergaard M, Benveniste H. Brain-wide pathway for waste clearance captured by contrast-enhanced MRI. J Clin Invest. 2013 Mar;123(3):1299-309. doi: 10.1172/JCI67677. Epub 2013 Feb 22. PMID 23434588
- [Background] Xavier ALR, Hauglund NL, von Holstein-Rathlou S, Li Q, Sanggaard S, Lou N, Lundgaard I, Nedergaard M. Cannula Implantation into the Cisterna Magna of Rodents. J Vis Exp. 2018 May 23;(135):57378. doi: 10.3791/57378. PMID 29889209
- [Background] Xie L, Kang H, Xu Q, Chen MJ, Liao Y, Thiyagarajan M, O'Donnell J, Christensen DJ, Nicholson C, Iliff JJ, Takano T, Deane R, Nedergaard M. Sleep drives metabolite clearance from the adult brain. Science. 2013 Oct 18;342(6156):373-7. doi: 10.1126/science.1241224. PMID 24136970
- [Background] Neely JD, Amiry-Moghaddam M, Ottersen OP, Froehner SC, Agre P, Adams ME. Syntrophin-dependent expression and localization of Aquaporin-4 water channel protein. Proc Natl Acad Sci U S A. 2001 Nov 20;98(24):14108-13. doi: 10.1073/pnas.241508198. PMID 11717465
- [Background] Munk AS, Wang W, Bechet NB, Eltanahy AM, Cheng AX, Sigurdsson B, Benraiss A, Mae MA, Kress BT, Kelley DH, Betsholtz C, Mollgard K, Meissner A, Nedergaard M, Lundgaard I. PDGF-B Is Required for Development of the Glymphatic System. Cell Rep. 2019 Mar 12;26(11):2955-2969.e3. doi: 10.1016/j.celrep.2019.02.050. PMID 30865886
- [Background] Amiry-Moghaddam M, Otsuka T, Hurn PD, Traystman RJ, Haug FM, Froehner SC, Adams ME, Neely JD, Agre P, Ottersen OP, Bhardwaj A. An alpha-syntrophin-dependent pool of AQP4 in astroglial end-feet confers bidirectional water flow between blood and brain. Proc Natl Acad Sci U S A. 2003 Feb 18;100(4):2106-11. doi: 10.1073/pnas.0437946100. Epub 2003 Feb 10. PMID 12578959
- [Background] Simon MJ, Wang MX, Murchison CF, Roese NE, Boespflug EL, Woltjer RL, Iliff JJ. Transcriptional network analysis of human astrocytic endfoot genes reveals region-specific associations with dementia status and tau pathology. Sci Rep. 2018 Aug 17;8(1):12389. doi: 10.1038/s41598-018-30779-x. PMID 30120299
- [Background] Frigeri A, Nicchia GP, Nico B, Quondamatteo F, Herken R, Roncali L, Svelto M. Aquaporin-4 deficiency in skeletal muscle and brain of dystrophic mdx mice. FASEB J. 2001 Jan;15(1):90-98. doi: 10.1096/fj.00-0260com. PMID 11149896
- [Background] Frigeri A, Nicchia GP, Verbavatz JM, Valenti G, Svelto M. Expression of aquaporin-4 in fast-twitch fibers of mammalian skeletal muscle. J Clin Invest. 1998 Aug 15;102(4):695-703. doi: 10.1172/JCI2545. PMID 9710437
- [Background] Nicchia GP, Rossi A, Mola MG, Pisani F, Stigliano C, Basco D, Mastrototaro M, Svelto M, Frigeri A. Higher order structure of aquaporin-4. Neuroscience. 2010 Jul 28;168(4):903-14. doi: 10.1016/j.neuroscience.2010.02.008. Epub 2010 Feb 11. PMID 20153404
- [Background] Neely JD, Christensen BM, Nielsen S, Agre P. Heterotetrameric composition of aquaporin-4 water channels. Biochemistry. 1999 Aug 24;38(34):11156-63. doi: 10.1021/bi990941s. PMID 10460172
- [Background] Crane JM, Bennett JL, Verkman AS. Live cell analysis of aquaporin-4 m1/m23 interactions and regulated orthogonal array assembly in glial cells. J Biol Chem. 2009 Dec 18;284(51):35850-60. doi: 10.1074/jbc.M109.071670. PMID 19843522
- [Background] Suzuki H, Nishikawa K, Hiroaki Y, Fujiyoshi Y. Formation of aquaporin-4 arrays is inhibited by palmitoylation of N-terminal cysteine residues. Biochim Biophys Acta. 2008 Apr;1778(4):1181-9. doi: 10.1016/j.bbamem.2007.12.007. Epub 2007 Dec 15. PMID 18179769
- [Background] Frigeri A, Gropper MA, Umenishi F, Kawashima M, Brown D, Verkman AS. Localization of MIWC and GLIP water channel homologs in neuromuscular, epithelial and glandular tissues. J Cell Sci. 1995 Sep;108 ( Pt 9):2993-3002. doi: 10.1242/jcs.108.9.2993. PMID 8537439
- [Background] Nagelhus EA, Mathiisen TM, Ottersen OP. Aquaporin-4 in the central nervous system: cellular and subcellular distribution and coexpression with KIR4.1. Neuroscience. 2004;129(4):905-13. doi: 10.1016/j.neuroscience.2004.08.053. PMID 15561407
- [Background] Jung JS, Bhat RV, Preston GM, Guggino WB, Baraban JM, Agre P. Molecular characterization of an aquaporin cDNA from brain: candidate osmoreceptor and regulator of water balance. Proc Natl Acad Sci U S A. 1994 Dec 20;91(26):13052-6. doi: 10.1073/pnas.91.26.13052. PMID 7528931
- [Background] Hasegawa H, Ma T, Skach W, Matthay MA, Verkman AS. Molecular cloning of a mercurial-insensitive water channel expressed in selected water-transporting tissues. J Biol Chem. 1994 Feb 25;269(8):5497-500. PMID 7509789
- [Background] Zakharov A, Papaiconomou C, Koh L, Djenic J, Bozanovic-Sosic R, Johnston M. Integrating the roles of extracranial lymphatics and intracranial veins in cerebrospinal fluid absorption in sheep. Microvasc Res. 2004 Jan;67(1):96-104. doi: 10.1016/j.mvr.2003.08.004. PMID 14709407
- [Background] McComb JG. Recent research into the nature of cerebrospinal fluid formation and absorption. J Neurosurg. 1983 Sep;59(3):369-83. doi: 10.3171/jns.1983.59.3.0369. PMID 6886750
- [Background] Upton ML, Weller RO. The morphology of cerebrospinal fluid drainage pathways in human arachnoid granulations. J Neurosurg. 1985 Dec;63(6):867-75. doi: 10.3171/jns.1985.63.6.0867. PMID 4056901
- [Background] Kido DK, Gomez DG, Pavese AM Jr, Potts DG. Human spinal arachnoid villi and granulations. Neuroradiology. 1976 Sep 21;11(5):221-8. doi: 10.1007/BF00328377. PMID 980235
- [Background] Mokri B. The Monro-Kellie hypothesis: applications in CSF volume depletion. Neurology. 2001 Jun 26;56(12):1746-8. doi: 10.1212/wnl.56.12.1746. PMID 11425944
- [Background] Sweetman B, Linninger AA. Cerebrospinal fluid flow dynamics in the central nervous system. Ann Biomed Eng. 2011 Jan;39(1):484-96. doi: 10.1007/s10439-010-0141-0. Epub 2010 Aug 25. PMID 20737291
- [Background] Zhu YC, Dufouil C, Soumare A, Mazoyer B, Chabriat H, Tzourio C. High degree of dilated Virchow-Robin spaces on MRI is associated with increased risk of dementia. J Alzheimers Dis. 2010;22(2):663-72. doi: 10.3233/JAD-2010-100378. PMID 20847444
- [Background] Potter GM, Chappell FM, Morris Z, Wardlaw JM. Cerebral perivascular spaces visible on magnetic resonance imaging: development of a qualitative rating scale and its observer reliability. Cerebrovasc Dis. 2015;39(3-4):224-31. doi: 10.1159/000375153. Epub 2015 Mar 19. PMID 25823458
- [Background] Wardlaw JM, Benveniste H, Nedergaard M, Zlokovic BV, Mestre H, Lee H, Doubal FN, Brown R, Ramirez J, MacIntosh BJ, Tannenbaum A, Ballerini L, Rungta RL, Boido D, Sweeney M, Montagne A, Charpak S, Joutel A, Smith KJ, Black SE; colleagues from the Fondation Leducq Transatlantic Network of Excellence on the Role of the Perivascular Space in Cerebral Small Vessel Disease. Perivascular spaces in the brain: anatomy, physiology and pathology. Nat Rev Neurol. 2020 Mar;16(3):137-153. doi: 10.1038/s41582-020-0312-z. Epub 2020 Feb 24. PMID 32094487
- [Background] Bechet NB, Shanbhag NC, Lundgaard I. Glymphatic pathways in the gyrencephalic brain. J Cereb Blood Flow Metab. 2021 Sep;41(9):2264-2279. doi: 10.1177/0271678X21996175. Epub 2021 Feb 27. PMID 33641515
- [Background] Ramos M, Burdon Bechet N, Battistella R, Pavan C, Xavier ALR, Nedergaard M, Lundgaard I. Cisterna Magna Injection in Rats to Study Glymphatic Function. Methods Mol Biol. 2019;1938:97-104. doi: 10.1007/978-1-4939-9068-9_7. PMID 30617975
- [Background] Bechet NB, Shanbhag NC, Lundgaard I. Direct Cannula Implantation in the Cisterna Magna of Pigs. J Vis Exp. 2021 Jun 9;(172). doi: 10.3791/62641. PMID 34180907
- [Background] Barshes N, Demopoulos A, Engelhard HH. Anatomy and physiology of the leptomeninges and CSF space. Cancer Treat Res. 2005;125:1-16. doi: 10.1007/0-387-24199-x_1. PMID 16211880
- [Background] Marques F, Sousa JC, Brito MA, Pahnke J, Santos C, Correia-Neves M, Palha JA. The choroid plexus in health and in disease: dialogues into and out of the brain. Neurobiol Dis. 2017 Nov;107:32-40. doi: 10.1016/j.nbd.2016.08.011. Epub 2016 Aug 18. PMID 27546055
- [Background] Spector R, Keep RF, Robert Snodgrass S, Smith QR, Johanson CE. A balanced view of choroid plexus structure and function: Focus on adult humans. Exp Neurol. 2015 May;267:78-86. doi: 10.1016/j.expneurol.2015.02.032. Epub 2015 Mar 4. PMID 25747036
- [Background] Ringstad G, Valnes LM, Dale AM, Pripp AH, Vatnehol SS, Emblem KE, Mardal KA, Eide PK. Brain-wide glymphatic enhancement and clearance in humans assessed with MRI. JCI Insight. 2018 Jul 12;3(13):e121537. doi: 10.1172/jci.insight.121537. PMID 29997300
- [Background] Eide PK, Ringstad G. MRI with intrathecal MRI gadolinium contrast medium administration: a possible method to assess glymphatic function in human brain. Acta Radiol Open. 2015 Nov 17;4(11):2058460115609635. doi: 10.1177/2058460115609635. eCollection 2015 Nov. PMID 26634147
- [Background] Nielsen S, Nagelhus EA, Amiry-Moghaddam M, Bourque C, Agre P, Ottersen OP. Specialized membrane domains for water transport in glial cells: high-resolution immunogold cytochemistry of aquaporin-4 in rat brain. J Neurosci. 1997 Jan 1;17(1):171-80. doi: 10.1523/JNEUROSCI.17-01-00171.1997. PMID 8987746
- [Background] Abbott NJ, Pizzo ME, Preston JE, Janigro D, Thorne RG. The role of brain barriers in fluid movement in the CNS: is there a 'glymphatic' system? Acta Neuropathol. 2018 Mar;135(3):387-407. doi: 10.1007/s00401-018-1812-4. Epub 2018 Feb 10. PMID 29428972
- [Background] Rennels ML, Gregory TF, Blaumanis OR, Fujimoto K, Grady PA. Evidence for a 'paravascular' fluid circulation in the mammalian central nervous system, provided by the rapid distribution of tracer protein throughout the brain from the subarachnoid space. Brain Res. 1985 Feb 4;326(1):47-63. doi: 10.1016/0006-8993(85)91383-6. PMID 3971148
- [Background] Groeschel S, Chong WK, Surtees R, Hanefeld F. Virchow-Robin spaces on magnetic resonance images: normative data, their dilatation, and a review of the literature. Neuroradiology. 2006 Oct;48(10):745-54. doi: 10.1007/s00234-006-0112-1. Epub 2006 Aug 5. PMID 16896908
- [Background] Dunker RO, Harris AB, Jenkins DP. Kinetics of horseradish peroxidase migration through cerebral cortex. Brain Res. 1976 Dec 17;118(2):199-217. doi: 10.1016/0006-8993(76)90708-3. PMID 1000288
- [Background] Oreskovic D, Klarica M, Vukic M. The formation and circulation of cerebrospinal fluid inside the cat brain ventricles: a fact or an illusion? Neurosci Lett. 2002 Jul 19;327(2):103-6. doi: 10.1016/s0304-3940(02)00395-6. PMID 12098646
- [Background] Bulat M, Lupret V, Orehkovic D, Klarica M. Transventricular and transpial absorption of cerebrospinal fluid into cerebral microvessels. Coll Antropol. 2008 Jan;32 Suppl 1:43-50. PMID 18405057
- [Background] Dandy WE. EXPERIMENTAL HYDROCEPHALUS. Ann Surg. 1919 Aug;70(2):129-42. doi: 10.1097/00000658-191908000-00001. No abstract available. PMID 17864139
- [Background] Dandy WE. INTRACRANIAL TUMORS AND ABSCESSES CAUSING COMMUNICATING HYDROCEPHALUS. Ann Surg. 1925 Aug;82(2):199-207. doi: 10.1097/00000658-192508000-00002. No abstract available. PMID 17865301
- [Background] Ahn JH, Cho H, Kim JH, Kim SH, Ham JS, Park I, Suh SH, Hong SP, Song JH, Hong YK, Jeong Y, Park SH, Koh GY. Meningeal lymphatic vessels at the skull base drain cerebrospinal fluid. Nature. 2019 Aug;572(7767):62-66. doi: 10.1038/s41586-019-1419-5. Epub 2019 Jul 24. PMID 31341278
- [Background] Weed LH. Studies on Cerebro-Spinal Fluid. No. IV : The dual Source of Cerebro-Spinal Fluid. J Med Res. 1914 Sep;31(1):93-118.11. No abstract available. PMID 19972195
- [Background] Mantovani G, Menegatti M, Scerrati A, Cavallo MA, De Bonis P. Controversies and Misconceptions Related to Cerebrospinal Fluid Circulation: A Review of the Literature from the Historical Pioneers' Theories to Current Models. Biomed Res Int. 2018 Nov 26;2018:2928378. doi: 10.1155/2018/2928378. eCollection 2018. PMID 30598991
- [Background] Zhou H, Andonegui G, Wong CH, Kubes P. Role of endothelial TLR4 for neutrophil recruitment into central nervous system microvessels in systemic inflammation. J Immunol. 2009 Oct 15;183(8):5244-50. doi: 10.4049/jimmunol.0901309. Epub 2009 Sep 28. PMID 19786543
- [Background] Rustenhoven J, Drieu A, Mamuladze T, de Lima KA, Dykstra T, Wall M, Papadopoulos Z, Kanamori M, Salvador AF, Baker W, Lemieux M, Da Mesquita S, Cugurra A, Fitzpatrick J, Sviben S, Kossina R, Bayguinov P, Townsend RR, Zhang Q, Erdmann-Gilmore P, Smirnov I, Lopes MB, Herz J, Kipnis J. Functional characterization of the dural sinuses as a neuroimmune interface. Cell. 2021 Feb 18;184(4):1000-1016.e27. doi: 10.1016/j.cell.2020.12.040. Epub 2021 Jan 27. PMID 33508229
- [Background] Karimy JK, Zhang J, Kurland DB, Theriault BC, Duran D, Stokum JA, Furey CG, Zhou X, Mansuri MS, Montejo J, Vera A, DiLuna ML, Delpire E, Alper SL, Gunel M, Gerzanich V, Medzhitov R, Simard JM, Kahle KT. Inflammation-dependent cerebrospinal fluid hypersecretion by the choroid plexus epithelium in posthemorrhagic hydrocephalus. Nat Med. 2017 Aug;23(8):997-1003. doi: 10.1038/nm.4361. Epub 2017 Jul 10. PMID 28692063
- [Background] Plog BA, Dashnaw ML, Hitomi E, Peng W, Liao Y, Lou N, Deane R, Nedergaard M. Biomarkers of traumatic injury are transported from brain to blood via the glymphatic system. J Neurosci. 2015 Jan 14;35(2):518-26. doi: 10.1523/JNEUROSCI.3742-14.2015. PMID 25589747
- [Background] Lavi E, Cong L. Type I astrocytes and microglia induce a cytokine response in an encephalitic murine coronavirus infection. Exp Mol Pathol. 2020 Aug;115:104474. doi: 10.1016/j.yexmp.2020.104474. Epub 2020 May 23. PMID 32454103
- [Background] Zhang R, Liu Y, Chen Y, Li Q, Marshall C, Wu T, Hu G, Xiao M. Aquaporin 4 deletion exacerbates brain impairments in a mouse model of chronic sleep disruption. CNS Neurosci Ther. 2020 Feb;26(2):228-239. doi: 10.1111/cns.13194. Epub 2019 Jul 31. PMID 31364823
- [Background] Rainey-Smith SR, Mazzucchelli GN, Villemagne VL, Brown BM, Porter T, Weinborn M, Bucks RS, Milicic L, Sohrabi HR, Taddei K, Ames D, Maruff P, Masters CL, Rowe CC, Salvado O, Martins RN, Laws SM; AIBL Research Group. Genetic variation in Aquaporin-4 moderates the relationship between sleep and brain Abeta-amyloid burden. Transl Psychiatry. 2018 Feb 26;8(1):47. doi: 10.1038/s41398-018-0094-x. PMID 29479071
- [Background] Wang LJ, Pan LN, Yan RY, Quan WW, Xu ZH. Obstructive sleep apnea increases heart rhythm disorders and worsens subsequent outcomes in elderly patients with subacute myocardial infarction. J Geriatr Cardiol. 2021 Jan 28;18(1):30-38. doi: 10.11909/j.issn.1671-5411.2021.01.002. PMID 33613657
- [Background] Spira AP, Gamaldo AA, An Y, Wu MN, Simonsick EM, Bilgel M, Zhou Y, Wong DF, Ferrucci L, Resnick SM. Self-reported sleep and beta-amyloid deposition in community-dwelling older adults. JAMA Neurol. 2013 Dec;70(12):1537-43. doi: 10.1001/jamaneurol.2013.4258. PMID 24145859
- [Background] Harrison IF, Ismail O, Machhada A, Colgan N, Ohene Y, Nahavandi P, Ahmed Z, Fisher A, Meftah S, Murray TK, Ottersen OP, Nagelhus EA, O'Neill MJ, Wells JA, Lythgoe MF. Impaired glymphatic function and clearance of tau in an Alzheimer's disease model. Brain. 2020 Aug 1;143(8):2576-2593. doi: 10.1093/brain/awaa179. PMID 32705145
- [Background] Iliff JJ, Chen MJ, Plog BA, Zeppenfeld DM, Soltero M, Yang L, Singh I, Deane R, Nedergaard M. Impairment of glymphatic pathway function promotes tau pathology after traumatic brain injury. J Neurosci. 2014 Dec 3;34(49):16180-93. doi: 10.1523/JNEUROSCI.3020-14.2014. PMID 25471560
- [Background] Taoka T, Naganawa S. Imaging for central nervous system (CNS) interstitial fluidopathy: disorders with impaired interstitial fluid dynamics. Jpn J Radiol. 2021 Jan;39(1):1-14. doi: 10.1007/s11604-020-01017-0. Epub 2020 Jul 11. PMID 32653987
- [Background] Agarwal N, Lewis LD, Hirschler L, Rivera LR, Naganawa S, Levendovszky SR, Ringstad G, Klarica M, Wardlaw J, Iadecola C, Hawkes C, Carare RO, Wells J, Bakker ENTP, Kurtcuoglu V, Bilston L, Nedergaard M, Mori Y, Stoodley M, Alperin N, de Leon M, van Osch MJP. Current Understanding of the Anatomy, Physiology, and Magnetic Resonance Imaging of Neurofluids: Update From the 2022 "ISMRM Imaging Neurofluids Study group" Workshop in Rome. J Magn Reson Imaging. 2024 Feb;59(2):431-449. doi: 10.1002/jmri.28759. Epub 2023 May 4. PMID 37141288
- [Background] Braun M, Iliff JJ. The impact of neurovascular, blood-brain barrier, and glymphatic dysfunction in neurodegenerative and metabolic diseases. Int Rev Neurobiol. 2020;154:413-436. doi: 10.1016/bs.irn.2020.02.006. Epub 2020 Jul 14. PMID 32739013
- [Background] Mestre H, Mori Y, Nedergaard M. The Brain's Glymphatic System: Current Controversies. Trends Neurosci. 2020 Jul;43(7):458-466. doi: 10.1016/j.tins.2020.04.003. Epub 2020 May 15. PMID 32423764
- [Background] Norwood JN, Zhang Q, Card D, Craine A, Ryan TM, Drew PJ. Anatomical basis and physiological role of cerebrospinal fluid transport through the murine cribriform plate. Elife. 2019 May 7;8:e44278. doi: 10.7554/eLife.44278. PMID 31063132
- [Background] Proulx ST. Cerebrospinal fluid outflow: a review of the historical and contemporary evidence for arachnoid villi, perineural routes, and dural lymphatics. Cell Mol Life Sci. 2021 Mar;78(6):2429-2457. doi: 10.1007/s00018-020-03706-5. Epub 2021 Jan 11. PMID 33427948
- [Background] Szentistvanyi I, Patlak CS, Ellis RA, Cserr HF. Drainage of interstitial fluid from different regions of rat brain. Am J Physiol. 1984 Jun;246(6 Pt 2):F835-44. doi: 10.1152/ajprenal.1984.246.6.F835. PMID 6742132
- [Background] Mestre H, Hablitz LM, Xavier AL, Feng W, Zou W, Pu T, Monai H, Murlidharan G, Castellanos Rivera RM, Simon MJ, Pike MM, Pla V, Du T, Kress BT, Wang X, Plog BA, Thrane AS, Lundgaard I, Abe Y, Yasui M, Thomas JH, Xiao M, Hirase H, Asokan A, Iliff JJ, Nedergaard M. Aquaporin-4-dependent glymphatic solute transport in the rodent brain. Elife. 2018 Dec 18;7:e40070. doi: 10.7554/eLife.40070. PMID 30561329
- [Background] DANDY WE. Treatment of an unusual subdural hydroma (external hydrocephalus). Arch Surg (1920). 1946 Apr;52:421-8. doi: 10.1001/archsurg.1946.01230050428003. No abstract available. PMID 20983109
- [Background] Weed LH. Studies on Cerebro-Spinal Fluid. No. III : The pathways of escape from the Subarachnoid Spaces with particular reference to the Arachnoid Villi. J Med Res. 1914 Sep;31(1):51-91. No abstract available. PMID 19972194
- [Background] Iliff JJ, Wang M, Liao Y, Plogg BA, Peng W, Gundersen GA, Benveniste H, Vates GE, Deane R, Goldman SA, Nagelhus EA, Nedergaard M. A paravascular pathway facilitates CSF flow through the brain parenchyma and the clearance of interstitial solutes, including amyloid beta. Sci Transl Med. 2012 Aug 15;4(147):147ra111. doi: 10.1126/scitranslmed.3003748. PMID 22896675
- [Background] Aspelund A, Antila S, Proulx ST, Karlsen TV, Karaman S, Detmar M, Wiig H, Alitalo K. A dural lymphatic vascular system that drains brain interstitial fluid and macromolecules. J Exp Med. 2015 Jun 29;212(7):991-9. doi: 10.1084/jem.20142290. Epub 2015 Jun 15. PMID 26077718
- [Background] Mazzitelli JA, Smyth LCD, Cross KA, Dykstra T, Sun J, Du S, Mamuladze T, Smirnov I, Rustenhoven J, Kipnis J. Cerebrospinal fluid regulates skull bone marrow niches via direct access through dural channels. Nat Neurosci. 2022 May;25(5):555-560. doi: 10.1038/s41593-022-01029-1. Epub 2022 Mar 17. PMID 35301477
- [Background] Suter T, Biollaz G, Gatto D, Bernasconi L, Herren T, Reith W, Fontana A. The brain as an immune privileged site: dendritic cells of the central nervous system inhibit T cell activation. Eur J Immunol. 2003 Nov;33(11):2998-3006. doi: 10.1002/eji.200323611. PMID 14579268
- [Background] Louveau A, Smirnov I, Keyes TJ, Eccles JD, Rouhani SJ, Peske JD, Derecki NC, Castle D, Mandell JW, Lee KS, Harris TH, Kipnis J. Structural and functional features of central nervous system lymphatic vessels. Nature. 2015 Jul 16;523(7560):337-41. doi: 10.1038/nature14432. Epub 2015 Jun 1. PMID 26030524
- [Background] Williams LR, Leggett RW. Reference values for resting blood flow to organs of man. Clin Phys Physiol Meas. 1989 Aug;10(3):187-217. doi: 10.1088/0143-0815/10/3/001. PMID 2697487
- [Background] Meng L, Hou W, Chui J, Han R, Gelb AW. Cardiac Output and Cerebral Blood Flow: The Integrated Regulation of Brain Perfusion in Adult Humans. Anesthesiology. 2015 Nov;123(5):1198-208. doi: 10.1097/ALN.0000000000000872. PMID 26402848
- [Background] Nedergaard M. Neuroscience. Garbage truck of the brain. Science. 2013 Jun 28;340(6140):1529-30. doi: 10.1126/science.1240514. PMID 23812703
- [Background] Jessen NA, Munk AS, Lundgaard I, Nedergaard M. The Glymphatic System: A Beginner's Guide. Neurochem Res. 2015 Dec;40(12):2583-99. doi: 10.1007/s11064-015-1581-6. Epub 2015 May 7. PMID 25947369
- [Result] Hattingen E, Jurcoane A, Melber J, Blasel S, Zanella FE, Neumann-Haefelin T, Singer OC. Diffusion tensor imaging in patients with adult chronic idiopathic hydrocephalus. Neurosurgery. 2010 May;66(5):917-24. doi: 10.1227/01.NEU.0000367801.35654.EC. PMID 20404696
- [Result] Ogata Y, Ozaki A, Ota M, Oka Y, Nishida N, Tabu H, Sato N, Hanakawa T. Interhemispheric Resting-State Functional Connectivity Predicts Severity of Idiopathic Normal Pressure Hydrocephalus. Front Neurosci. 2017 Sep 1;11:470. doi: 10.3389/fnins.2017.00470. eCollection 2017. PMID 28919849
- [Result] Leinonen V, Menon LG, Carroll RS, Dello Iacono D, Grevet J, Jaaskelainen JE, Black PM. Cerebrospinal fluid biomarkers in idiopathic normal pressure hydrocephalus. Int J Alzheimers Dis. 2011;2011:312526. doi: 10.4061/2011/312526. Epub 2011 Jun 1. PMID 21660204